CLINICAL TRIAL: NCT04797494
Title: A Randomized Controlled Trial On Testing A New Vertical Dimension Of Occlusion Prior To Restorative Treatment Of Generalized Tooth Wear
Brief Title: Testing New Vertical Dimension Of Occlusion Prior To Restorative Treatment Of Tooth Wear
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL31371.091.10
Record Dates: First submitted 2021-03-08; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Tooth Wear; Randomized Controlled Trial; Vertical Dimension of Occlusion; Composite Resins
Keywords: Randomized controlled trial; Rehabilitation
MeSH Terms: conditions — Tooth Wear

STUDY DESIGN:
Intervention Model Description: This study is a Randomized Controlled Trial (RCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): No acrylic Removable Appliance (RA) was prescribed for patients prior to restorative treatment of generalized severe tooth wear.
- Experimental Group (Experimental): A acrylic Removable Appliance (RA) was prescribed for patients prior to restorative treatment of generalized severe tooth wear. Patients were asked to wear the RA 3 weeks prior to restorative treatment for 24h per day, except for when eating.
  Interventions: Device: acrylic removable appliance

INTERVENTIONS:
Device: acrylic removable appliance — Hand-made, dental laboratory-manufactured, acrylic removable appliances were made on the mandible after intraoral impressions (Alginate, Cavex).
  Patients were asked to wear the RA for a period of 3 weeks prior to restorative treatment, for 24 h per day, except for when eating.
  Arms: Experimental Group

SUMMARY:
This study is a Randomized Controlled Trial (RCT). The aim of the study is to evaluate the necessity to test the desired increased Vertical Dimension of Occlusion (VDO) prior to restorative treatment of generalized tooth wear.

Tooth wear is a physiological phenomenon, that when becoming pathological, can result in functional problems such as pain, reduced quality of life and esthetic impairment. Restorative treatment should be discussed with patients with severe or pathological tooth wear.

The restorative treatment of generalized tooth wear includes restoration of teeth, separately, in increased VDO. The increment of VDO is based upon clinical parameters such as the amount of natural tooth tissue, the possibility to lengthen the anterior teeth in regard to an acceptable esthetics outcome, and the Free Way Space (FWS). The FWS is the intermaxillary space when the masticatory-muscles-complex is relaxed.

Traditionally, it is believed that adapting to a new VDO results in clinical difficulties such as different speech, pain of the Temporo Mandibular Joint (TMJ), masticatory muscle pain, and increased masticatory muscles activity. The latter could result in an increased bite force and (possibly) an increased failure rate of restorations. Some operators, then, prefer to test the increment of VDO prior to restorative treatment to check if patients can adjust to the new VDO. This raises the question if the needed increment of VDO to restore worn dentitions should be checked prior to restorative treatment. The hypothesis in this study is that testing the needed increment of VDO prior to restorative treatment does not improve the restorative treatment.

Patients with generalized severe tooth wear were included and restoratively treated with composite restorations. Prior to restorative treatment, patients were randomized to either receiving an acrylic Removable Appliance (RA) or no RA. The RA was worn for 3 weeks prior to restorative treatment and included the intended increment of VDO. These patients were asked to wear the RA during the whole day, except when eating.

After restorative treatment, patients revisited our dental clinic after 1 month and after 1 year. Quality of life was assessed with questionnaires. FWS was assessed clinically. Restorations were checked for clinical acceptability, including small materials fractures.

DETAILED DESCRIPTION:
This study is a Randomized Controlled Trial (RCT). The aim of the study is to evaluate the necessity to test the increased Vertical Dimension of Occlusion (VDO) prior to restorative treatment of generalized tooth wear.

Tooth wear is a physiological phenomenon, that when becoming pathological, can result in functional problems such as pain, reduced quality of life and esthetic impairment. Restorative treatment should be discussed in with patients with severe or pathological tooth wear.

The restorative treatment includes restoration of all teeth, separately, in increased VDO. The increment of VDO is based upon clinical parameters as the amount of loss of natural tooth tissue, the possibility to lengthen the maxillary anterior teeth in regard to an acceptable esthetic outcome, and the Free Way Space (FWS). The FWS is the intermaxillary space when the masticatory-muscles-complex is relaxed.

Traditionally, it is believed that adapting to a new VDO results in clinical difficulties such as different speech, pain of the Temporo Mandibular Joint (TMJ), masticatory muscle pain, and increased masticatory muscles activity. The latter could result in an increased bite force and an increased failure rate of restorations. Some operators, then, prefer to test the increment of VDO prior to restorative treatment to check if patients can adjust to the new VDO. This raises the question if the needed increment of VDO to restore worn dentitions should be checked prior to restorative treatment. The hypothesis in this study is that testing the needed increment of VDO prior to restorative treatment does not improve the adaptation to the restorative treatment.

The research was registered in the ClinicalTrial.gov register after the study had been completed. This RCT is part of RCT with a 2x2 design. The first branch was used to randomize patients to certain restorative protocol, which was enlisted in ClinicalTrials.gov (NCT04326816). The second branch was designed to test the VDO prior to restorative treatment of generalized severe tooth wear. Approval of the local Medical-Ethics-committee (METC) for the 2x2 RCT was sought and granted in 2010. Approval was granted to a protocol in which no Data Safety Monitoring Board was appointed as research standards were different in 2010. The study was conducted according to the principles of the Declaration of Helsinki and in accordance with the Medical Research Involving Human Subjects Act (WMO).

Sample size calculation base done by a biostatistician. Calculations were completed based upon the first branch of the 2x2 RCT. A group size of 75 patients was established. Anonymized paper case report forms were completed at each moment and stored. A separate digital database was made and used for data analysis. Data analysis consisted of descriptive analysis of failed restorations and paired t-Test with a significance level of 5%. Serious Adverse Events (SAE) report files and Suspected Unexpected Serious Adverse Reaction (SUSAR) report files were present and could be, when necessary, filled in and applied to the local METC.

Patients were recruited as General Dental Practitioners (GDP) referred patients with generalized tooth wear to the academic clinic. Patients were seen by 1 operator and were assessed for eligibility. Patients received a written informed consent and were included if the informed consent was signed. Patients received an identification number C1 to C49. A randomization was performed on the use of a removable appliance to test the VDO prior to restorative treatment. Randomization with a block size of eight was performed. The random sequence was put into envelopes. The investigator opened the envelope in their numbered order and assigned the patient to the corresponding group immediately after the consent was acquired.

A laboratory-made acrylic Removable Appliance (RA) was evaluated to test the adaptation of the patient to the increment of VDO. In the control group, no RA was prescribed prior to restorative treatment. In the test group, a RA was prescribed prior to restorative treatment. Patients were asked to wear the RA for 24h per day, with the exception for when eating, during a period of 3 weeks. Thereafter, the acceptance was checked using a questionnaire.

Data collection was done at predetermined moments i.e., baseline, immediately after treatment, 1 month after treatment, 1 year after treatment. During the recall moments, Oral Health-related Quality of Life (OHRQoL) was assessed using questionnaires, as was the FWS. In addition, restorations were checked based on clinical acceptability and all failures were recorded.

No specific Quality assurance plan to address data validation and registry procedures, including site monitoring and auditing was made prior to the onset of the study.

Data checks were completed by 1 researcher. Source data verification to assess the accuracy, completeness, and representativeness was completed by 1 researcher. Medical records (Electronic patient files), digital photos made at recall appointments, and paper case report forms were inspected. No specific source data verification plan was made prior to the onset of the study.

ELIGIBILITY:
Inclusion Criteria:

* Generalized moderate to severe tooth wear with patient demand for treatment
* Full dental arches, one diastema due to one missing posterior tooth was allowed
* Estimated need for an increase in VDO of at least 3 mm in the first molar region

Exclusion Criteria:

* Limited mouth opening
* (History of) Temporomandibular dysfunction
* Advanced periodontitis, deep caries lesions, or multiple large restorations including teeth with endodontic problems

Patients with specific individual risk factors, such as parafunctional habits of grinding/clenching or patients with Gastro-Oesophageal Reflux Disease (GORD), were not excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2016-02-14 (Actual); Study Completion 2016-02-14 (Actual)

PRIMARY OUTCOMES:
Interventions on restorations | Baseline, recall after 1 month, recall after 1 year.
  Number of interventions needed for patients to adjust to the increased VDO

SECONDARY OUTCOMES:
Oral Health Impact Profile (OHIP) questionnaire | Baseline, Recall after 1 month, recall after 1 year.
  To assess the Oral Health-related Quality of Life (OHRQoL), OHIP questionnaires were completed by patients at different moments. The questionnaire consists of 46 specific questions which can be scored on a 1 to 5 ordinal scale. Higher scores mean a worse outcome.
Orofacial Esthetic Scale (OES) questionnaire | Baseline, Recall after 1 month, recall after 1 year.
  To assess the Oral Health-related Quality of Life (OHRQoL), OES questionnaires were completed by patients at different moments. The questionnaire used an 11-point ordinal scale, ranging from very dissatisfied (0) to very satisfied (10). It consisted of 8 questions. Item 1 to 7 addressed the appearance of the face, profile, mouth, tooth alignment, tooth shape, tooth color, and gums. The last item (8) characterizes the patient's overall assessment of orofacial esthetics. Higher scores mean a better outcome.
Free Way Space | Baseline, Recall after 1 month, recall after 1 year.
  The space between the occluding surfaces of the maxillary and mandibular

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Charlotte Huysmans, Prof. Dr., Study Chair — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No